CLINICAL TRIAL: NCT01573481
Title: Pressure Controlled Ventilation Versus Pressure Support Ventilation During the Night: New Strategy of Mechanical Ventilation Weaning?
Brief Title: Comparison of Two Ventilator Mode During the Night: New Strategy of Mechanical Ventilation Weaning
Acronym: REVENTIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI2012_843_0016
Record Dates: First submitted 2012-02-22; First posted 2012-04-09 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Weaning Failure; COPD Exacerbation
Keywords: WEANING; PRESSURE CONTROLLED CONTINOUS VENTILATION; PRESSURE VENTILATION SUPPORT; SLEEP; POLYGRAPHIC RECORD

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure support ventilation (Active Comparator): Patients in this group are ventilated during the night (10 PM to 9 AM) with pressure support ventilation mode. The level of the pressure support is the same as the previous day.
  During the day (9 AM to 10 PM), patients are ventilated with pressure support ventilation (the level of pressure support is progressively decreased).
  Interventions: Other: pressure support ventilation
- Pressure controlled ventilation (Active Comparator): Patients in this group are ventilated during the night (10 PM to 9 AM) with pressure controlled ventilation mode. The level of inspiratory pressure is set to 20 cm H2O and the respiratory rate is adjusted to avoid any spontaneous breathing (respiratory rate > or equal to 12 breath per min). During the day (9 AM to 10 PM), patients are ventilated with pressure support ventilation (the level of pressure support is progressively decreased).
  Interventions: Other: Pressure controlled ventilation

INTERVENTIONS:
Other: pressure support ventilation — Patients in this group are ventilated during the night with pressure support ventilation mode. The level of the pressure support is the same as the previous day.
  Arms: Pressure support ventilation
Other: Pressure controlled ventilation — Patients in this group are ventilated during the night (10 PM to 9 AM) with pressure controlled ventilation mode. The level of inspiratory pressure is set to 20 cm H2O and the respiratory rate is adjusted to avoid any spontaneous breathing (respiratory rate > or equal to 12 breath per min).
  Arms: Pressure controlled ventilation

SUMMARY:
The purpose of the study is to compare pressure controlled continuous mandatory ventilation versus pressure support ventilation during the night for weaning to mechanical ventilation in chronic obstructive pulmonary disease patients and their impact onto sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* The patient and/or legal representative of the patient has provided a written informed consent before inclusion in the study
* The patients is hospitalized in respiratory and critical care unit (university hospital of AMIENS, FRANCE)
* the patient is mechanically ventilated (ventilator model : puritan-bennett B840)
* Pulmonary disease,chronic obstructive (Spirometry and Blood Gas Analysis in chronic state before admission)
* stable cardiovascular status (cardiac frequency < 140 beats/min and systolic blood pressure : 90-160 mmHg without catecholamines)
* midazolam < 0,05mg/kg/h
* sufentanyl < 0,05µ/kg/h
* the disorder that caused respiratory failure and prompted mechanical ventilation is treated
* the clinician suspects the patient may be ready to begin the weaning process
* inspiratory oxygen fraction (FiO2) < 50%
* positive end-expiratory pressure < or equal 8cmH2O
* during the day, the patient tolerate pressure support ventilation (pressure support level < 15cmH2O
* respiratory frequency (FR) < 35 breaths/min
* tidal volume (VT) > 5ml/kg
* PaO2/FiO2 > 200 mmHg
* FR/VT < 105 breaths/min/L

Exclusion Criteria:

* sleep apnea, central
* narcolepsy
* Encephalopathy, Metabolic AND Encephalitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Weaning duration | between one to 21 days (the study will begin when patient presents weaning criteria and will stop 48 days after extubation.)
  weaning duration in days (from the first day with spontaneous ventilation to extubation)

SECONDARY OUTCOMES:
weaning failure | 48 hours
  Failure of weaning = re-intubation, necessity of non invative ventilation support for periods during the day time or death, in the first 48 hours following extubation
Quantity and quality of sleep | 1 to 21 days
  Polygraphic datas will be analyzed during weaning, integrating: Proportion of sleep stages (I, II, III, IV, REM sleep), overall sleep and awakeness period.
  Average ratio of diurnal sleep on total overall sleep, average ratio of diurnal sleep on total sleep at the first day of weaning and the day before extubation; Observation of central apneas from begining of weaning to extubation.

CONTACTS AND LOCATIONS:
Overall Officials: ANDREJAK Claire, MD, Principal Investigator — CHU Amiens; JOUNIEAUX Vincent, MD PhD, Study Director — CHU Amiens; BASILLE Damien, MD, Principal Investigator — CHU Amiens; ROGER Pierre-Alexandre, MD, Principal Investigator — CHU Amiens; ROSE Dominique, MD, Principal Investigator — CHU Amiens; MONCONDUIT Julien, MD, Principal Investigator — CHU Amiens
Locations (1):
- Pneumologie et Réanimation Respiratoire, Amiens, France

REFERENCES:
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Epstein SK, Ciubotaru RL, Wong JB. Effect of failed extubation on the outcome of mechanical ventilation. Chest. 1997 Jul;112(1):186-92. doi: 10.1378/chest.112.1.186. PMID 9228375
- [Background] Brochard L, Rauss A, Benito S, Conti G, Mancebo J, Rekik N, Gasparetto A, Lemaire F. Comparison of three methods of gradual withdrawal from ventilatory support during weaning from mechanical ventilation. Am J Respir Crit Care Med. 1994 Oct;150(4):896-903. doi: 10.1164/ajrccm.150.4.7921460.
- [Background] Esteban A, Frutos F, Tobin MJ, Alia I, Solsona JF, Valverdu I, Fernandez R, de la Cal MA, Benito S, Tomas R, et al. A comparison of four methods of weaning patients from mechanical ventilation. Spanish Lung Failure Collaborative Group. N Engl J Med. 1995 Feb 9;332(6):345-50. doi: 10.1056/NEJM199502093320601. PMID 7823995
- [Background] Esteban A, Alia I. Clinical management of weaning from mechanical ventilation. Intensive Care Med. 1998 Oct;24(10):999-1008. doi: 10.1007/s001340050708. No abstract available. PMID 9840232
- [Background] Aurell J, Elmqvist D. Sleep in the surgical intensive care unit: continuous polygraphic recording of sleep in nine patients receiving postoperative care. Br Med J (Clin Res Ed). 1985 Apr 6;290(6474):1029-32. doi: 10.1136/bmj.290.6474.1029. PMID 3921096
- [Background] Hilton BA. Quantity and quality of patients' sleep and sleep-disturbing factors in a respiratory intensive care unit. J Adv Nurs. 1976 Nov;1(6):453-68. doi: 10.1111/j.1365-2648.1976.tb00932.x. No abstract available. PMID 1050357
- [Background] Freedman NS, Gazendam J, Levan L, Pack AI, Schwab RJ. Abnormal sleep/wake cycles and the effect of environmental noise on sleep disruption in the intensive care unit. Am J Respir Crit Care Med. 2001 Feb;163(2):451-7. doi: 10.1164/ajrccm.163.2.9912128. PMID 11179121
- [Background] Schwab RJ. Disturbances of sleep in the intensive care unit. Crit Care Clin. 1994 Oct;10(4):681-94. PMID 8000921
- [Background] Parthasarathy S, Tobin MJ. Effect of ventilator mode on sleep quality in critically ill patients. Am J Respir Crit Care Med. 2002 Dec 1;166(11):1423-9. doi: 10.1164/rccm.200209-999OC. Epub 2002 Sep 5. PMID 12406837
- [Background] Parreira VF, Delguste P, Jounieaux V, Aubert G, Dury M, Rodenstein DO. Effectiveness of controlled and spontaneous modes in nasal two-level positive pressure ventilation in awake and asleep normal subjects. Chest. 1997 Nov 5;112(5):1267-77. doi: 10.1378/chest.112.5.1267. PMID 9367467
- [Background] Parreira VF, Delguste P, Jounieaux V, Aubert G, Dury M, Rodenstein DO. Glottic aperture and effective minute ventilation during nasal two-level positive pressure ventilation in spontaneous mode. Am J Respir Crit Care Med. 1996 Dec;154(6 Pt 1):1857-63. doi: 10.1164/ajrccm.154.6.8970381.
- [Background] Bosma K, Ferreyra G, Ambrogio C, Pasero D, Mirabella L, Braghiroli A, Appendini L, Mascia L, Ranieri VM. Patient-ventilator interaction and sleep in mechanically ventilated patients: pressure support versus proportional assist ventilation. Crit Care Med. 2007 Apr;35(4):1048-54. doi: 10.1097/01.CCM.0000260055.64235.7C. PMID 17334259
- [Background] Toublanc B, Rose D, Glerant JC, Francois G, Mayeux I, Rodenstein D, Jounieaux V. Assist-control ventilation vs. low levels of pressure support ventilation on sleep quality in intubated ICU patients. Intensive Care Med. 2007 Jul;33(7):1148-1154. doi: 10.1007/s00134-007-0659-2. Epub 2007 May 11. PMID 17492431
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. PMID 8254858
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Teasdale G, Murray G, Parker L, Jennett B. Adding up the Glasgow Coma Score. Acta Neurochir Suppl (Wien). 1979;28(1):13-6. doi: 10.1007/978-3-7091-4088-8_2. No abstract available. PMID 290137
- [Background] Riker RR, Picard JT, Fraser GL. Prospective evaluation of the Sedation-Agitation Scale for adult critically ill patients. Crit Care Med. 1999 Jul;27(7):1325-9. doi: 10.1097/00003246-199907000-00022. PMID 10446827
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Hansen-Flaschen J, Cowen J, Polomano RC. Beyond the Ramsay scale: need for a validated measure of sedating drug efficacy in the intensive care unit. Crit Care Med. 1994 May;22(5):732-3. No abstract available. PMID 8181279
- [Result] Andrejak C, Monconduit J, Rose D, Toublanc B, Mayeux I, Rodenstein D, Jounieaux V. Does using pressure-controlled ventilation to rest respiratory muscles improve sleep in ICU patients? Respir Med. 2013 Apr;107(4):534-41. doi: 10.1016/j.rmed.2012.12.012. Epub 2013 Feb 4. PMID 23391488